CLINICAL TRIAL: NCT05887895
Title: A Trial Comparing the Pharmacodynamics and Pharmacokinetics of HR20014, INS068 and INS062 in Healthy Subjects
Brief Title: To Compare the Pharmacokinetics and Pharmacodynamics of HR20014, INS068 and INS062 After Single Subcutaneous Injection in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HR20014-102
Record Dates: First submitted 2023-05-08; First posted 2023-06-05 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: The study was a single-center, randomized, open, six-sequence, three-cycle crossover phase I study in healthy subjects. The objective of this trial was to compare the PK/PD and safety of HR20014, INS068 and INS062 in a single subcutaneous injection of the same dose.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Treatment group sequence 1 (Experimental): Subjects were given HR20014, INS068, or INS062 injections subcutaneously once in three cycles. The interval of each dosing visit was 7 to 21 days.
  Interventions: Drug: INS062 injection、INS068 injection、HR20014 injection
- Treatment group sequence 2 (Experimental): Subjects were given HR20014, INS062, or INS068 injections subcutaneously once in three cycles. The interval of each dosing visit was 7 to 21 days.
  Interventions: Drug: INS062 injection、INS068 injection、HR20014 injection
- Treatment group sequence 3 (Experimental): Subjects were given INS068, HR20014, or INS062 injections subcutaneously once in three cycles. The interval of each dosing visit was 7 to 21 days.
  Interventions: Drug: INS062 injection、INS068 injection、HR20014 injection
- Treatment group sequence 4 (Experimental): Subjects were given INS068, INS062, or HR20014 injections subcutaneously once in three cycles. The interval of each dosing visit was 7 to 21 days.
  Interventions: Drug: INS062 injection、INS068 injection、HR20014 injection
- Treatment group sequence 5 (Experimental): Subjects were given INS062, HR20014, or INS068 injections subcutaneously once in three cycles. The interval of each dosing visit was 7 to 21 days.
  Interventions: Drug: INS062 injection、INS068 injection、HR20014 injection
- Treatment group sequence 6 (Experimental): Subjects were given INS062, INS068, or HR20014 injections subcutaneously once in three cycles. The interval of each dosing visit was 7 to 21 days.
  Interventions: Drug: INS062 injection、INS068 injection、HR20014 injection

INTERVENTIONS:
Drug: INS062 injection、INS068 injection、HR20014 injection — INS062 injection：A single dose of 0.4 DU/kg is administered to healthy subjects.
  INS068 injection：A single dose of 0.4 U/kg is administered to healthy subjects.
  HR20014 injection：A single dose of 0.4 U/kg is administered to healthy subjects.

SUMMARY:
This is a single-center, randomized, open, six-sequence, three-period crossover phase I clinical trial in healthy subjects to compare the PK/PD and safety profiles of single dose of HR20014, INS068, and INS062. In this study, 12 subjects were randomly assigned to 6 administration sequences in a ratio of 1:1:1:1:1:1, and HR20014, INS068 or INS062 injection were given subcutaneously three times before and after each sequence.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent;
2. Male or female aged 18-45 at screening (both inclusive);
3. Subjects who are considered to be generally healthy, based on an assessment of medical history, physical examination and clinical laboratory data, as judged by the Investigator;
4. Male weight ≥ 50.0 kg, female weight ≥ 45.0 kg, body mass index (BMI) in 18.0~26.0 kg/m2 (both inclusive);
5. During the screening phase oral glucose tolerance test (OGTT), intravenous fasting plasma glucose ≥3.9 mmol/L and < 6.1 mmol/L; Glucose 2 hours after negative charge static pulse blood sugar <7.8mmol/L； and normal or abnormal insulin levels have no clinical significance.

Exclusion Criteria:

1. A history of recurrent or severe drug food allergy, or known or suspected allergy to any component of the study drug;
2. Have a history of hypertension;
3. Severe systemic infectious diseases within 1 month before screening;
4. Patients with a history of lower extremity deep vein thrombosis or high risk of lower extremity deep vein thrombosis;
5. Patients with serious diseases of the psychiatric, cardiovascular, respiratory, digestive, endocrine, blood, urogenital and other systems in the past, or existing diseases of the above systems, were judged by the researchers to be unfit to participate in this study;
6. Use of prescription drugs (topical eye/nasal drops and creams and occasional antipyretic and analgesic drugs such as acetaminophen within recommended doses are permitted) and over-the-counter drugs, and Chinese herbal medicine (regular vitamins are allowed) within 2 weeks before screening;
7. Presence of any abnormal and clinically significant laboratory tests.
8. ECG (12-lead electrocardiogram) showed abnormal and clinically significant.
9. Those who have participated in any drug clinical trials within 3 months or 5 half-life periods before screening (the elder shall prevail), who participated in clinical trials are defined as random, prior to screening.
10. Blood donation within 1 month before screening; Or patients with trauma or major surgical procedures who donated blood or lost blood ≥400 mL in the 3 months prior to screening.
11. Women who are pregnant, breastfeeding or planning to conceive, or women of childbearing potential (WOCBP) are reluctant to use appropriate contraception during the trial.
12. The investigators determined that other conditions were inappropriate for participation in this clinical trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-07-18 (Actual)

PRIMARY OUTCOMES:
Area under the Glucose Infusion Rate (GIR) - time curve (Only for HR20014 and INS068） | 0 hour to 6 hours after dosing
Area under the Glucose Infusion Rate (GIR) - time curve (Only for HR20014 and INS062） | 6 hours to 24 hours after dosing

SECONDARY OUTCOMES:
Area under the Glucose Infusion Rate (GIR) - time curve | 0 hour to 96 hours after dosing
  Based on the absolute dose and concentration of INS068
Maximum concentration of INS068 | 0 hour to 96 hours after dosing
  Based on the absolute dose and concentration of INS068
Area under the Glucose Infusion Rate (GIR) - time curve | 0 hour to 10 hours after dosing
  Based on the absolute dose and concentration of INS062
Maximum concentration of INS062 | 0 hour to 10 hours after dosing
  Based on the absolute dose and concentration of INS062
Incidence and severity of adverse events (AEs) | from screening to 7-21 days after the last dosing

CONTACTS AND LOCATIONS:
Locations (1):
- The second affiliated hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided